CLINICAL TRIAL: NCT01422148
Title: Minocycline Plus Amiodarone Versus Amiodarone Alone for the Prevention of Atrial Fibrillation After Cardiac Surgery (MINA)
Brief Title: Minocycline Plus Amiodarone Versus Amiodarone Alone for the Prevention of Atrial Fibrillation After Cardiac Surgery
Acronym: MINA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Responsible Party: Principal Investigator, Abdallah Alameddine, Medical Staff, Baystate Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BH-09-176
Record Dates: First submitted 2011-08-17; First posted 2011-08-23 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation
Keywords: cardiac surgery; atrial fibrillation; minocycline; amiodarone
MeSH Terms: conditions — Atrial Fibrillation; cyclopia sequence | interventions — Amiodarone; Minocycline

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Amiodarone (Other): oral amiodarone
  Interventions: Drug: Amiodarone
- minocycline (Experimental): intravenous minocycline 100 mg daily x 5 days starting intra-operatively combined with oral amiodarone (400 mg twice daily for 7 days, then 200 mg twice daily for the next 7 days
  Interventions: Drug: Amiodarone; Drug: Minocycline

INTERVENTIONS:
Drug: Amiodarone — oral amiodarone (400 mg twice daily for 7 days, then 200 mg twice daily for the next 7 days
Drug: Minocycline — intravenous minocycline 100 mg daily x 5 days starting intra-operatively combined with oral amiodarone (400 mg twice daily for 7 days, then 200 mg twice daily for the next 7 days
  Other Names: Minocin
  Arms: minocycline

SUMMARY:
. New- onset postoperative atrial fibrillation (POAF) is a common complication after cardiac surgery and its occurrence increases with age. POAF can result in clinically significant morbidity and mortality. The national trend in the US is that the population older than 65 years is increasing, making healthcare expenditure related to POAF to be a major burden on health care system. Effective treatment of POAF is imperative in ensuring quality of care and reduction of costs.

In 2021 there is a projected total of 377,763 cardiovascular surgeries in the US alone with approximately half of which will have POAF with longer postoperative length of stay (+3.9 days) and higher discharge costs (+$13,993) than no-POAF patients (Reference: Ann Thorac Surg. 2015 Jan;99(1):109-14). Amiodarone, the currently used therapy, is often insufficient to prevent POAF and has multiple side-effects. In this study, we expect to improve the incidence of POAF by using a common acne drug (Minocycline) that is safe and that could be incorporated in clinical care of this disease.

DETAILED DESCRIPTION:
New-onset postoperative atrial fibrillation after cardiac surgery (POAF) is commonly observed and it increases morbidity, mortality, and health care expenditure. Amiodarone administration is proposed initial agent for prevention and treatment of POAF, but while useful, this drug has a number of adverse side-effects and relapse requiring anticoagulation therapy at hospital discharge is prevalent. Effective medications are needed with respect to management. Minocycline, an old tetracycline antibiotic, has additional effects including inhibition of atrial myocyte apoptosis.The finding that apoptosis of right atrial myocytes is thought to be one etiologic factor underlying POAF supports examining the hypothesis in this project that adding minocycline to amiodarone could favorably reduce POAF frequency rate. Minocycline has been used for over four decades and has a good safety profile, therefore this investigation is not a phase I trial. With a limited sample size, while the data of our MINAA Exploratory trial (the Minocycline Plus Amiodarone Versus Amiodarone Alone for the Prevention of Atrial Fibrillation After Cardiac Surgery) were not sufficient to draw definite conclusions, rather they suggested feasibility of such therapy in this cohort. In the current pilot study, we assess the clinical effectiveness and safety of minocycline plus amiodarone in preventing POAF with a larger cohort of two parallel groups (n=40, each) randomly assigned in a 1:1 ratio.In this trial we compare intravenous minocycline 100 mg daily x 5 days starting intra-operatively combined with oral amiodarone (400 mg twice daily for 7 days, then 200 mg twice daily for the next 7 days), versus the same dose oral amiodarone alone, for prevention of POAF among adult patients undergoing coronary artery bypass grafts, heart valve repair or replacement, or combined procedures. All patients receive 150 mg intravenous amiodarone intraoperatively and a 2nd similar dose of amiodarone bolus is permitted for tachyarrhythmia any time within 24 hours after surgery.The primary outcome is a newly detected POAF by telemetry, Holter monitoring, or by daily wireless ECG sensors within 6 weeks from the time of randomization. Composite secondary outcomes include death at 30 days, length of hospital stay, and other adverse events.To elucidate how minocycline causally elicits its pharmacologic effects, sera sampling of biomarkers such as NF-Kappa B, cleaved caspase-3, and NT-pro-BNP are measured pre-procedure, then on the 3rd and 5th postoperative days. If the proposed intervention is successful, it underscores what can ensue when the target evolves to the common population level requiring a nuanced approach pursued by Phase III-IV proposals

ELIGIBILITY:
Inclusion criteria are adults, including women and minorities > 18 years of age, who are also willing to participate for the duration of the trial (6 weeks). All non-congenital cardiac operations are included: Coronary Artery Bypass Graft, valve repair/replacement, or combination of CABG and heart valve operations. Patients should be able to access iPhones and download ECGs using their electronic Devices. Exclusion criteria Patients with prior (within 6 months) or current atrial fibrillation (AF) or flutter, patients undergoing concomitant surgical AF ablation or a history of AF, transcatheter aortic valve replacement or other minimally invasive procedures, prior cerebrovascular event, cardiogenic shock or resuscitation, evidence of hepatic or renal dysfunctions (i.e., an alanine aminotransferase level that is ≥ twice the upper limit of the normal range, or either a serum creatinine level that is ≥ 2.0 mg/dL or need for preoperative dialysis) are excluded. Other exclusion criteria are the following: thyrotoxicosis, pregnancy, severe chronic obstructive pulmonary disease (COPD, with FEV1/FVC <70%), recent history of drug or alcohol abuse, and intolerance to tetracycline or amiodarone. Because a core scientific basis of this trial concerning the role of underlying atrial tissue inflammatory/apoptotic activity, patients with inflammatory conditions such as lupus, severe arthritis, thyroiditis or inflammatory bowel disease are excluded; as are patients taking preoperative immunosuppressant agents, long-term (>10 days) oral corticosteroids (prednisolone > 10mg or other), or estrogen replacement; and finally patients with newly diagnosed cancer (<5 years) are also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-01-24 (Estimated); Study Completion 2028-01-24 (Estimated)

PRIMARY OUTCOMES:
Post-op Atrial Fibrillation | 6 weeks
  frequency of a newly detected episode of POAF occuring after the initial surgery, or within 6 weeks after hospital discharge

SECONDARY OUTCOMES:
Thromboembolism | 6 weeks
  cerebral or pulmonary
Heart failure | 6 weeks
  Symptoms include dyspnea, leg edema, low Ejection Fraction, high Central Venous Pressure, high level of natriuretic hormone
30-day hospital death | 30-days
  cardiac or overall

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah k Alameddine, MD, Principal Investigator — Baystate Medical Center
Locations (1):
- Abdallah Alameddine, Melrose, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Three years
Access Criteria: de-identified computerized dataset